CLINICAL TRIAL: NCT03390400
Title: Intraindividual Comparison of Prostaglandin E2 (PGE2) and Total-prostaglandin (PG) Following Femtosecond Laser-assisted Cataract Surgery Using a Low-energy, High-frequency Femtosecond Laser-Device in Regard to the Sequence of Anterior Capsulotomy and Lens Fragmentation
Brief Title: Changes in Prostaglandin Levels in Laser Cataract Surgery (LCS) Subject to Laser Prevalence
Acronym: Femto-PG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rupert Menapace (Other)
Responsible Party: Sponsor-Investigator, Rupert Menapace, Prof. Dr. med. univ., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Femto-PGII Study
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Age Related Cataracts
Keywords: Laser Cataract Surgery

STUDY DESIGN:
Intervention Model Description: Bilateral femtosecond-laser assisted cataract surgery will be performed in individuals with age-related cataract. Eyes will be randomized into two groups receiving either anterior capsulotomy before lens fragmentation or vice versa in the contralateral eye. After laser procedure samples of aqueous humor will be collected and when complete all samples will be analysed by ELISA for Prostaglandin.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Groups will be randomized. Randomization information will be put in a sealed envelope on screening date and opened in operating theatre right before procedure start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Capsulotomy before Lens Fragmentation (Active Comparator): Anterior capsulotomy will be performed by femtosecond laser before lens fragmentation
  Interventions: Device: Femtosecondlaser-assisted; Procedure: Anterior Capsulotomy
- Lens Fragmentation before Anterior Capsulotomy (Active Comparator): Lens fragmentation will be performed by femtosecond laser before anterior capsulotomy
  Interventions: Device: Femtosecondlaser-assisted; Procedure: Lens Fragmentation

INTERVENTIONS:
Device: Femtosecondlaser-assisted — Femtosecondlaser-assisted Cataract Surgery will be performed bilateral on the same day with different laser settings.
  Other Names: Laser assisted Cataract Surgery
Procedure: Anterior Capsulotomy — Cataract Surgery
  Arms: Anterior Capsulotomy before Lens Fragmentation
Procedure: Lens Fragmentation — Cataract Surgery
  Arms: Lens Fragmentation before Anterior Capsulotomy

SUMMARY:
The investigational device is an approved femtosecond laser (FSL) device with an integrated imaging system to perform certain steps of the cataract procedure. The FSL will perform anterior capsulotomy and lens fragmentation in individuals suffering from age-related cataract with need of cataract surgery.

Cataract surgery will be performed in subjects who have signed an informed consent form. Aqueous humor will be collected and screening will be performed for Total Prostaglandin and Prostaglandin E2 via en-bloc Enzyme-linked Immunosorbent Assay (ELISA)-Kit.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract necessitating phacoemulsification extraction and posterior intraocular lens implantation
* Age: 40 to 90 (females of childbearing age will be interviewed if pregnancy is possible)
* Preoperative pupil dilation in mydriasis ≥ 6.5 mm

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Recurrent intraocular inflammation of unknown etiology
* Uncontrolled glaucoma
* Uncontrolled systemic or ocular disease
* Blind fellow eye
* Microphthalmus
* Corneal abnormality
* History of uveitis/iritis
* Iris neovascularization
* Pseudoexfoliation
* Proliferative diabetic retinopathy
* Pregnancy
* Lactation
* Females of childbearing age: not included

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-03-14 (Estimated)

PRIMARY OUTCOMES:
Total-Prostaglandin and PGE2 level in aqueous humor | 5 minutes after laser procedure (LCS)
  pg/mL

SECONDARY OUTCOMES:
Change in Pupilsize | baseline, immediately after laser, 5 min after laser
  in mm

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No